CLINICAL TRIAL: NCT07360093
Title: Evaluation of the Clinical Effectiveness of Pericapsular Nerve Group (PENG) Block and Pulsed Radiofrequency Applications in Chronic Hip Pain
Acronym: PENG-PRF
Status: Not yet recruiting | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Ülkü Sabuncu, Assoc. Prof., Ankara City Hospital Bilkent
Other Study IDs: 123456
Record Dates: First submitted 2026-01-14; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Osteoarthritis (OA) of the Hip
Keywords: Osteoarthritis, Hip,; Pain, Chronic; Nerve Blockade; Pulsed Radiofrequency Treatment
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Hip; Chronic Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group PENG: The initial step in patients diagnosed with chronic hip pain is a diagnostic intervention, namely the application of a pericapsular nerve group (PENG) block. In patients who benefit from the diagnostic block-defined as a reduction of 50% or more in VAS scores following the procedure-pulsed radiofrequency (PRF) treatment is added as a second-stage intervention. This stepwise approach reflects our standard clinical practice, and both procedures are commonly used in our clinic for the management of chronic hip pain. However, the available evidence in the literature on this approach is largely limited to case reports and retrospective case series. The aim of the present study is to document and share the clinical outcomes of this treatment strategy that we routinely apply in clinical practice.
  Interventions: Procedure: PENG Block Pulsed radiofrequency

INTERVENTIONS:
Procedure: PENG Block Pulsed radiofrequency — This intervention consists of a stepwise, two-stage treatment protocol routinely applied in our clinical practice for the management of chronic hip pain. In the first stage, all patients undergo an ultrasound-guided pericapsular nerve group (PENG) block as a diagnostic and therapeutic procedure. Pain intensity is assessed using the Visual Analog Scale (VAS) following the diagnostic block. Only patients who demonstrate a clinically meaningful response, defined as a reduction of 50% or greater in VAS scores, proceed to the second stage of the intervention.
  In the second stage, pulsed radiofrequency (PRF) treatment is applied to the same target region in addition to the PENG block, aiming to achieve longer-lasting analgesia through neuromodulation without tissue destruction. All procedures are performed under ultrasound guidance by experienced pain specialists using standardized techniques. This stepwise, response-guided combination approach distinguishes the present intervention from si

SUMMARY:
The primary aim of this study is to prospectively compare the effects of the pericapsular nerve group (PENG) block alone and the combination of PENG block with pulsed radiofrequency (PRF) on pain intensity in patients with chronic hip pain. As a secondary aim, the effects of both treatment modalities on hip function are intended to be evaluated using valid and reliable functional assessment scales. Through this study, it is aimed to demonstrate the clinical contribution of adding PRF to the PENG block and to identify a more effective and longer-lasting approach for the interventional treatment of chronic hip pain.

DETAILED DESCRIPTION:
Chronic hip pain is a common clinical condition, particularly in the elderly, that significantly impairs quality of life and leads to functional limitation and dependence in daily activities. Chronic hip pain caused by degenerative, inflammatory, and mechanical conditions-most notably hip osteoarthritis-often remains inadequately controlled despite medical treatment, physical therapy, and rehabilitation. Although surgical interventions can be effective, they are not suitable for all patients due to advanced age, comorbidities, or surgical contraindications. Therefore, minimally invasive interventional pain management techniques have gained increasing importance in the treatment of chronic hip pain.

The nociceptive innervation of the hip joint primarily arises from the anterior capsule, which is mainly supplied by the sensory branches of the femoral, obturator, and accessory obturator nerves. Based on this anatomical rationale, the pericapsular nerve group (PENG) block is an ultrasound-guided technique that targets these sensory fibers to provide effective analgesia without causing motor blockade. Previous studies have shown that the PENG block reduces pain scores and improves functional mobility in both acute and chronic hip pain; however, its analgesic effect may be time-limited, requiring repeated applications in some patients.

Pulsed radiofrequency (PRF), unlike conventional thermal radiofrequency, aims to modulate nerve transmission without causing tissue destruction and may provide longer-lasting analgesia through neuromodulatory mechanisms. Recent evidence suggests that combining PRF with peripheral nerve blocks may prolong analgesic effects compared with nerve blocks alone. However, prospective studies directly comparing PENG block alone with PENG block combined with PRF in chronic hip pain are limited, highlighting the need for further investigation.

ELIGIBILITY:
Inclusion Criteria:

* Presence of chronic hip pain lasting at least 3 months

Baseline Visual Analog Scale (VAS) score ≥ 4

Clinical and/or radiological diagnosis of hip osteoarthritis or non-specific chronic hip pain

Inadequate response to conservative treatments

Written informed consent obtained

Exclusion Criteria:

* Local or systemic infection at the intervention site

Coagulopathy or inability to discontinue anticoagulant therapy

Hip pain related to malignancy

History of previous hip arthroplasty

Severe neurological deficit

Pregnancy or breastfeeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 18-80 years old with chronical hip pain
Sampling Method: Non-Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Primary outcome | baseline (pre-procedure) and at 1 week, 1 month, 3 months, and 6 months after the procedure.
  NRS: numeric rating scale

SECONDARY OUTCOMES:
Secondary outcome | baseline (pre-procedure) and at 1 week, 1 month, 3 months, and 6 months after the procedure.
  WOMAC score: Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC).
  Harris Hip Score: hip function evaluation

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] 10.5152/TJAR.2021.21230